CLINICAL TRIAL: NCT05723107
Title: Phase I Pilot Study of Endoscopic Ultrasound Guided RFA in Advanced Pancreatic Cancer
Brief Title: EUS RFA for Treatment of Pancreatic Ductal Adenocarcinoma (PDAC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Taewoong Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-00249
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Chemotherapy plus EUS-RFA (Experimental): Endoscopic ultrasound-guided radiofrequency ablation (EUS-RFA) and chemotherapy will be administered as part of standard of care treatment for PDAC in patients receiving palliative second- or third-line therapy for unresectable non-metastatic pancreatic cancer.
  Study participants will undergo 3 identical EUS-RFA procedures, administered during Study Window 2 (Weeks 1-3), Window 3 (Weeks 5-7), and Window 4 (Weeks 9-11). During each EUS-RFA procedure, a tumor biopsy will also be taken for single cell RNA sequencing.
  Chemotherapy will be administered during Study Window 2 (Weeks 1-3), Window 3 (Weeks 5-7), Window 4 (Weeks 9-11), and Window 5 (Weeks 13-15).
  Interventions: Drug: Chemotherapy; Device: Endoscopic Ultrasound-Guided Radiofrequency Ablation (EUS-RFA)

INTERVENTIONS:
Drug: Chemotherapy — Patients will receive continuation of second or initiate third-line chemotherapy regimen at the discretion and decision of treating oncologist.
Device: Endoscopic Ultrasound-Guided Radiofrequency Ablation (EUS-RFA) — EUS-RFA will be delivered using the EUSRA RF Electrode, which is a sterile, single-use electrosurgical accessory for coagulation and ablation of soft tissue when used in conjunction with compatible radio frequency generator (VIVA Combo RF Generator).
  The device will be used during a routine EUS, which is a minimally invasive procedure used to assess gastrointestinal diseases. Each EUS-RFA procedure will last approximately 60 minutes.
  Other Names: EUSRA RF Electrode

SUMMARY:
This is a single arm study in the treatment of pancreatic ductal adenocarcinoma (PDAC). The investigators propose to test the tolerability of chemotherapy plus endoscopic ultrasound-guided radiofrequency ablation (EUS-RFA) using the RF Electrode in patients receiving palliative second or third line therapy for unresectable non-metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and histologically confirmed PDAC by biopsy
* Axial CT scan or MRI consistent with PDAC with at least 1 cm in greatest diameter
* ECOG performance status 0-2
* Patients with locally advanced PDAC, who have not responded or progressed on first line chemotherapy, are deemed not resectable based on multidisciplinary review, and show no evidence of distant metastasis
* Lesions between 1 - 4cm in size

Exclusion Criteria:

* Patients that show evidence of distant metastasis
* Endoscopically non-accessible mass
* Pregnant patients
* Inability to provide informed consent
* Lesions <1cm, or >4cm in greatest diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Complete Therapy without Grade III-IV Adverse Events (AEs) as Assessed by CTCAE v. 5.0 | Up to Week 15
  Per Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0, Grade III AEs are defined as severe or medically significant but not immediately life-threatening; or hospitalization or prolongation of hospitalization indicated; or disabling; or limiting self care activities of daily living. Grade IV AEs are defined as life-threatening consequences; or urgent intervention indicated.

SECONDARY OUTCOMES:
Percentage of Participants who Complete all 3 EUS-RFA Treatments | Up to Week 11
  Treatments delivered during Study Window 2 (Weeks 1-3), Window 3 (Weeks 5-7), and Window 4 (Weeks 9-11).
Disease-Free Survival from Diagnosis | Up to Week 24
  Time from diagnosis to first clinical evidence of local or distant recurrence.
Disease-Free Survival from First Study Procedure | Up to Week 24
  Time from first study procedure (delivered during Weeks 1-3) to first clinical evidence of local or distant recurrence.
Overall Survival From Diagnosis | Up to Week 24
  Time from diagnosis to death.
Percentage of Participants who Report Post-Procedural Complications | Up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Tamas A. Gonda, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Tisch Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Tamas.Gonda@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Tamas.Gonda@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.